CLINICAL TRIAL: NCT03530358
Title: MOdularity for SEnsory Motor Control: Implications of Muscle Synergies in Motor Recovery After Stroke
Brief Title: MOdularity for SEnsory Motor Control
Acronym: MOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Andrea Turolla, PT, PhD, IRCCS San Camillo, Venezia, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015.14; 16/GR-2011-02348942 (Other Grant/Funding Number: Ministero della Salute, Italy)
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Stroke, Ischemic; Upper Limb Injury; Rehabilitation
Keywords: Muscle Synergies; MRI; Virtual Reality; Robotics
MeSH Terms: conditions — Ischemic Stroke; Arm Injuries

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: A simple random number sequence will be generated by a computer and the allocation concealment will be guaranteed using sequentially numbered, opaque sealed envelopes. The therapists responsible for randomization and allocation procedures will be independent of the blind therapists and medical doctors involved in patients' screening and treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-aided rehabilitation (Experimental): The technology-aided upper limb rehabilitation include reinforced feedback in virtual environment (RFVE), or robotic therapy.
  Interventions: Device: Technology-aided rehabilitation
- Conventional rehabilitation (Active Comparator): The conventional upper limb rehabilitation program will be based on traditional rehabilitation techniques aimed at restoring upper limb motor functions.
  Interventions: Behavioral: Conventional rehabilitation

INTERVENTIONS:
Device: Technology-aided rehabilitation — VRRS involves performing different kinds of motor tasks with the patient holding a real manipulable object in their hands while interacting with a virtual scenario.
  "Braccio di Ferro" task consists in center-out reaching movements and return. The subject is required to start from a central target, reach one of five peripheral targets arranged on a semi-circle with a 20 cm radius and then return to the central target.
  Other Names: Virtual Reality Rehabilitation System (VRRS); Braccio di Ferro
  Arms: Technology-aided rehabilitation
Behavioral: Conventional rehabilitation — The patients will be asked to perform a wide range of exercises, including: shoulder flexion-extension, abduction-adduction, internal-external rotation, circumduction, elbow flexion-extension, forearm pronation-supination, hand-digit motion. Standardized instructions and modalities will be followed when providing exercises to the patients in order to control for any variability in leading the therapy session due to the therapist.
  Arms: Conventional rehabilitation

SUMMARY:
For this project the investigators ask, how the activation and organization of muscle synergies may be disrupted by brain lesions, and whether it is possible to modify synergy activations by means of specific therapies. Will be investigated whether there is a relationship between post-stroke cortical plasticity and changes in synergy activations due to a therapy.

DETAILED DESCRIPTION:
It has been widely recognized that neurorehabilitation can facilitate recovery of motor function after stroke. There has been increasing evidence suggesting that the execution of voluntary movement relies critically on the functional integration of the motor areas and the spinal circuitries. More precisely, it was suggested that the central nervous system may generate neural motor commands through a linear combination of spinal modules, each of which activates a group of muscles as a single unit (muscle synergy). The investigators hypothesize that descending motor cortical signals generate movements by combining and activating muscle synergies. With this background, the goal is to further improve the efficacy of rehabilitation utilizing knowledge on modular motor control. The investigators also seek to provide a better understanding of the links between brain activations and movements.

The project MO-SE has three aims, one primary and two secondary. The main primary aim is to test whether the use of virtual reality rehabilitation based therapies are superior in terms of clinical efficacy to conventional therapies (randomized clinica trial, RCT). The other two secondary aims of the project will be accomplished with further instrumental analysis in sub-samples of the group of patients enrolled for the RCT.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of first stroke;
* a score between 1 and 3 (included) at the upper limb sub-item on the Italian version of the National Institute of Health stroke scale (IT - NIHSS) (Pezzella et al., 2009)
* a score higher than 6 out of 66 on the Fugl - Meyer upper extremity (F-M UE) scale (Fugl-Meyer et al., 1975).

Exclusion Criteria:

* the presence of a moderate cognitive decline defined as a Mini Mental State Examination (Folstein et al., 1975) score < 20/30 points;
* the finding of severe verbal comprehension deficit defined as a number of errors > 13 (Tau Points < 58/78) on the Token Test (Huber et al., 1984);
* evidence of apraxia and visuospatial neglect interfering with upper arm movements and manipulation of simple objects in all the directions within the visual field, as assessed through neurological examination;
* report in the patient's clinical history or evidence from the neurological examination of behavioural disturbances (i.e. delusions, aggressiveness and severe apathy/depression) that could affect compliance with the rehabilitation programs;
* non stabilised fractures;
* diagnosis of depression/delusion;
* associated traumatic brain injury;
* drug resistant epilepsy;
* evidence of ideomotor apraxia;
* evidence of visuospatial neglect;
* severe impairment of verbal comprehension defined as a score higher than 13 errors on Token test (i.e. score<58 out of 78 Tau points).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2014-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Scale - Upper Extremity (construct: upper limb motor function) | 20 days
  Scale range scores: 0 - 66 points. Total summed score is reported with higher values representing a better outcome.

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) (construct: measure for independence in the activities of daily living - ADLs) | 20 days
  Scale range scores: 18 - 126 points. Total summed score is reported with higher values representing a better outcome.
Fugl-Meyer Assessment Scale - Range of Motion of Joints (construct: measure joints' passive range of motion) | 20 days
  Scale range scores: 0 - 44 points. Total summed score is reported with higher values representing a better outcome.
Fugl-Meyer Assessment Scale - Sensory Function (construct: measure of residual sensory function in upper and lower limbs affected by paresis) | 20 days
  Scale range scores: 0 - 24 points. Total summed score is reported with higher values representing a better outcome.
Fugl-Meyer Assessment Scale - Balance (construct: measure of impairment of standing and balance functions) | 20 days
  Scale range scores: 0 - 14 points. Total summed score is reported with higher values representing a better outcome.
Reaching Performance Scale (construct: measure of the ability to reach targets in the frontal space of upper limb affected by paresis) | 20 days
  Scale range scores: 0 - 36 points. Total summed score is reported with higher values representing a better outcome.
Modified Ashworth Scale (construct: measure of spasticity at the upper limb) | 20 days
  Scale range scores: 0 - 5 ranks. Total summed ranks are reported with higher values representing a worse outcome.
Box and Block Test | 20 days
  Measure of gross motor function of the hand and upper limb

OTHER OUTCOMES:
Mean duration [s] | 20 days
  Time needed to execute standard motor tasks
Mean velocity [cm/s] | 20 days
  Velocity expressed to execute standard motor tasks
Smoothness [number of submovements] | 20 days
  Smoothness expressed to execute standard motor tasks
Muscle synergies [n] | 20 days
  Number of muscular patterns recognised by processing of surface electromyography data to execute standard motor tasks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Turolla, PhD, Principal Investigator — IRCCS San Camillo, Venezia, Italy
Locations (2):
- Italy (2):
  - IRCCS Fondazione Don Gnocchi Onlus, Milan
  - IRCCS San Camillo, Venezia, Italy, Venice

REFERENCES:
- [Background] Saltiel P, Wyler-Duda K, D'Avella A, Tresch MC, Bizzi E. Muscle synergies encoded within the spinal cord: evidence from focal intraspinal NMDA iontophoresis in the frog. J Neurophysiol. 2001 Feb;85(2):605-19. doi: 10.1152/jn.2001.85.2.605. PMID 11160497
- [Background] d'Avella A, Portone A, Fernandez L, Lacquaniti F. Control of fast-reaching movements by muscle synergy combinations. J Neurosci. 2006 Jul 26;26(30):7791-810. doi: 10.1523/JNEUROSCI.0830-06.2006. PMID 16870725
- [Background] Weiss T, Miltner WH, Liepert J, Meissner W, Taub E. Rapid functional plasticity in the primary somatomotor cortex and perceptual changes after nerve block. Eur J Neurosci. 2004 Dec;20(12):3413-23. doi: 10.1111/j.1460-9568.2004.03790.x. PMID 15610174
- [Background] Cheung VC, Piron L, Agostini M, Silvoni S, Turolla A, Bizzi E. Stability of muscle synergies for voluntary actions after cortical stroke in humans. Proc Natl Acad Sci U S A. 2009 Nov 17;106(46):19563-8. doi: 10.1073/pnas.0910114106. Epub 2009 Oct 30. PMID 19880747
- [Background] Cheung VC, Turolla A, Agostini M, Silvoni S, Bennis C, Kasi P, Paganoni S, Bonato P, Bizzi E. Muscle synergy patterns as physiological markers of motor cortical damage. Proc Natl Acad Sci U S A. 2012 Sep 4;109(36):14652-6. doi: 10.1073/pnas.1212056109. Epub 2012 Aug 20. PMID 22908288
- [Background] Mehrholz J, Hadrich A, Platz T, Kugler J, Pohl M. Electromechanical and robot-assisted arm training for improving generic activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD006876. doi: 10.1002/14651858.CD006876.pub3. PMID 22696362
- [Background] Laver KE, George S, Thomas S, Deutsch JE, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD008349. doi: 10.1002/14651858.CD008349.pub2. PMID 21901720
- [Background] Carpinella I, Cattaneo D, Abuarqub S, Ferrarin M. Robot-based rehabilitation of the upper limbs in multiple sclerosis: feasibility and preliminary results. J Rehabil Med. 2009 Nov;41(12):966-70. doi: 10.2340/16501977-0401. PMID 19841825
- [Background] Carpinella I, Cattaneo D, Bertoni R, Ferrarin M. Robot training of upper limb in multiple sclerosis: comparing protocols with or without manipulative task components. IEEE Trans Neural Syst Rehabil Eng. 2012 May;20(3):351-60. doi: 10.1109/TNSRE.2012.2187462. PMID 22623407
- [Background] Sacco RL, Wolf PA, Bharucha NE, Meeks SL, Kannel WB, Charette LJ, McNamara PM, Palmer EP, D'Agostino R. Subarachnoid and intracerebral hemorrhage: natural history, prognosis, and precursive factors in the Framingham Study. Neurology. 1984 Jul;34(7):847-54. doi: 10.1212/wnl.34.7.847. PMID 6539860
- [Background] Pezzella FR, Picconi O, De Luca A, Lyden PD, Fiorelli M. Development of the Italian version of the National Institutes of Health Stroke Scale: It-NIHSS. Stroke. 2009 Jul;40(7):2557-9. doi: 10.1161/STROKEAHA.108.534495. Epub 2009 Jun 11. PMID 19520997
- [Background] Keith RA, Granger CV, Hamilton BB, Sherwin FS. The functional independence measure: a new tool for rehabilitation. Adv Clin Rehabil. 1987;1:6-18. No abstract available. PMID 3503663
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Huber W, Poeck K, Willmes K. The Aachen Aphasia Test. Adv Neurol. 1984;42:291-303. No abstract available. PMID 6209953
- [Background] Lee DD, Seung HS. Learning the parts of objects by non-negative matrix factorization. Nature. 1999 Oct 21;401(6755):788-91. doi: 10.1038/44565. PMID 10548103
- [Background] Inzitari D, Carlucci G. Italian Stroke Guidelines (SPREAD): evidence and clinical practice. Neurol Sci. 2006 Jun;27 Suppl 3:S225-7. doi: 10.1007/s10072-006-0622-y. PMID 16752053
- [Background] Bamford J, Sandercock P, Dennis M, Burn J, Warlow C. Classification and natural history of clinically identifiable subtypes of cerebral infarction. Lancet. 1991 Jun 22;337(8756):1521-6. doi: 10.1016/0140-6736(91)93206-o. PMID 1675378
- [Background] Arya KN, Verma R, Garg RK. Estimating the minimal clinically important difference of an upper extremity recovery measure in subacute stroke patients. Top Stroke Rehabil. 2011 Oct;18 Suppl 1:599-610. doi: 10.1310/tsr18s01-599. PMID 22120029
- [Background] Piron L, Turolla A, Agostini M, Zucconi C, Tonin P, Piccione F, Dam M. Assessment and treatment of the upper limb by means of virtual reality in post-stroke patients. Stud Health Technol Inform. 2009;145:55-62. PMID 19592786
- [Background] Piron L, Turolla A, Agostini M, Zucconi CS, Ventura L, Tonin P, Dam M. Motor learning principles for rehabilitation: a pilot randomized controlled study in poststroke patients. Neurorehabil Neural Repair. 2010 Jul-Aug;24(6):501-8. doi: 10.1177/1545968310362672. PMID 20581337
- [Background] Basteris A, De Luca A, Sanguineti V, Solaro C, Mueller M, Carpinella I, Cattaneo D, Bertoni R, Ferrarin M. A tailored exercise of manipulation of virtual tools to treat upper limb impairment in Multiple Sclerosis. IEEE Int Conf Rehabil Robot. 2011;2011:5975509. doi: 10.1109/ICORR.2011.5975509. PMID 22275705
- [Background] Casadio M, Sanguineti V, Morasso PG, Arrichiello V. Braccio di Ferro: a new haptic workstation for neuromotor rehabilitation. Technol Health Care. 2006;14(3):123-42. PMID 16971753
- [Background] Bohannon RW, Andrews AW. Interrater reliability of hand-held dynamometry. Phys Ther. 1987 Jun;67(6):931-3. doi: 10.1093/ptj/67.6.931. PMID 3588679
- [Result] Lencioni T, Fornia L, Bowman T, Marzegan A, Caronni A, Turolla A, Jonsdottir J, Carpinella I, Ferrarin M. A randomized controlled trial on the effects induced by robot-assisted and usual-care rehabilitation on upper limb muscle synergies in post-stroke subjects. Sci Rep. 2021 Mar 5;11(1):5323. doi: 10.1038/s41598-021-84536-8. PMID 33674675
- [Result] Cheung VC, Devarajan K, Severini G, Turolla A, Bonato P. Decomposing time series data by a non-negative matrix factorization algorithm with temporally constrained coefficients. Annu Int Conf IEEE Eng Med Biol Soc. 2015 Aug;2015:3496-9. doi: 10.1109/EMBC.2015.7319146. PMID 26737046
- [Result] Turolla A, Venneri A, Farina D, Cagnin A, Cheung VCK. Rehabilitation Induced Neural Plasticity after Acquired Brain Injury. Neural Plast. 2018 May 10;2018:6565418. doi: 10.1155/2018/6565418. eCollection 2018. No abstract available. PMID 29861717
- [Derived] Carpinella I, Lencioni T, Bowman T, Bertoni R, Turolla A, Ferrarin M, Jonsdottir J. Effects of robot therapy on upper body kinematics and arm function in persons post stroke: a pilot randomized controlled trial. J Neuroeng Rehabil. 2020 Jan 30;17(1):10. doi: 10.1186/s12984-020-0646-1. PMID 32000790